CLINICAL TRIAL: NCT00442078
Title: Evaluation of the Efficacy on Urinary Continence and Quality of Life of the Sub-urethral Tape I-STOP® Using the Transobturator and Perineal Route on Male Incontinent After Radical Prostatectomy.
Brief Title: I-STOP TOMS - Trans Obturator Male Sling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CL Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020402
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Male Urinary Incontinence
Keywords: Incontinence; Urinary; Male; Tape; Transobturator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: I-STOP TOMS male sling — Bulbus urethral compression with polypropylene mesh

SUMMARY:
The main objective is to evaluate the clinical efficacy on continence, quality of life and tolerance of the sub-urethral tape I-STOP on male patient suffering of incontinence significant and embarrassing after a radical prostatectomy.

DETAILED DESCRIPTION:
Title

Evaluation of the efficacy on urinary continence and quality of life of the sub-urethral tape I-STOP using the transobturator and perineal route on male incontinent after radical prostatectomy.

Chief Investigator:

Pr. Philippe GRISE - Professor and Chairman of Urology Hopital Charles Nicolle, 1 rue de Germont, 76000 Rouen-FRANCE Tel+ 33.(0)2.32.88.81.73 Fax+ 33.(0)2.32.88.82.05 Email philippe.grise@chu-rouen.fr

Promoter Vincent GORIA - CEO CL Médical, 28, avenue Général de Gaulle, 69110 Sainte Foy Les Lyon - FRANCE Tel+33.(0)4.78.59.54.93 Fax+33.(0)4.78.59.89.78 Email vgoria@clmedical.com

Associate investigators

Forty urologist surgeons are involved on this study.

Objective

The main objective is to evaluate the clinical efficacy on continence, quality of life and tolerance of the sub-urethral tape I-STOP on male patient suffering of incontinence significant and embarrassing after a radical prostatectomy.

Methodology

Opened study, prospective, multicenter, with direct individual benefit.

Number of patients

50 patient minimum, with 1 to 3 patients for each investigator.

Duration Including: 12 months Follow-up: 12 months Total: 24 months

Key words Incontinence Urinary Male Tape Transobturator

ELIGIBILITY:
Inclusion Criteria:

* Male, with post-prostatectomy urinary incontinence (either after radical prostatectomy or prostatectomy of prostate adenoma, whatever the route used), and for whom there has been more than 6 months follow-up since the date of that procedure.
* The patient should have been proposed urinary re-education, which was refused for personal reasons, or should still suffer from urinary incontinence despite the re-education.
* Urinary incontinence is materialized in this population by a score between 4 and 16 (inclusive) for the three questions of the ICIQ questionnaire.
* A urodynamic assessment including flow measurement and residue will have been carried out.
* A urethroscopy or urethrography will have been carried out to eliminate cases of urethral stenosis.
* Inclusion is subject to obtaining informed written consent, after remittance of the information sheet, and having had a detailed medical examination carried out.
* Medication for urinary incontinence and in particular anticholinergic drugs must have been stopped at least 15 days prior to initial assessment and for the duration of the trial. The same goes for urinary re-education.

Exclusion Criteria:

* Progressing prostatic neoplasia materialized by testing of PSA levels.
* Prostate radiotherapy.
* Neurological disorder which might lead to urinary incontinence or hinder assessment.
* Urethral or anastomotic stenosis materialized by urethroscopy or urethrography.
* Hyperactive detrusor muscle with leakage contemporaneous with uninhibited contractility.
* Chronic retention of urine with leakage due to overflow.
* Current urinary infection. This would be a temporary exclusion since assessment can take place after treatment and monitoring for sterility of urine.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of continence and QoL with questionnaires and PAD test | 1 month, 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
UCLA SF36 score and ICIQ continence | 1-3-6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRISE, Professor, Principal Investigator — Rouen University Hospital - France
Locations (1):
- Rouen University Hospital, Rouen, France